CLINICAL TRIAL: NCT00709904
Title: A Multinational, Multicenter, Randomized, Double-Blind Study Comparing the Efficacy and Safety of AVE5026 With Placebo for the Extended Prevention of Venous Thromboembolism in Patients Having Undergone Hip Fracture Surgery
Brief Title: Evaluation of AVE5026 as Compared to Placebo for the Extended Prophylaxis of Venous Thromboembolism in Patients Having Undergone Hip Fracture Surgery
Acronym: SAVE-HIP3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EFC10636; 2007-007947-28 (EudraCT Number)
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-06

CONDITIONS: Venous Thromboembolism
Keywords: venous thromboprophylaxis; primary prevention; orthopedic surgery
MeSH Terms: conditions — Venous Thromboembolism | interventions — AVE 5026

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Semuloparin extension treatment (Experimental): Extension treatment with Semuloparin sodium 20 mg (10 mg if SRI) for 19-23 days following initial treatment with open-label Semuloparin 20 mg (10 mg if SRI) for 7-10 days.
  Interventions: Drug: Open-label Semuloparin sodium; Drug: Semuloparin sodium
- Placebo extension treatment (Placebo Comparator): Extension treatment with placebo (for Semuloparin sodium) for 19-23 days following initial treatment with open-label Semuloparin 20 mg (10 mg if SRI) for 7-10 days
  Interventions: Drug: Open-label Semuloparin sodium; Drug: Placebo (for Semuloparin sodium)

INTERVENTIONS:
Drug: Open-label Semuloparin sodium — 0.4 mL (0.2 mL if SRI) solution in ready-to-use 0.5 ml pre-filled syringe
  Subcutaneous injection once daily with an initial dose given 8 hours after surgery
  Other Names: AVE5026
Drug: Placebo (for Semuloparin sodium) — 0.4 mL (0.2 mL if SRI) solution in ready-to-use 0.5 ml prefilled syringe strictly identical in appearance containing the same volume but without active component
  Subcutaneous injection once daily
  Arms: Placebo extension treatment
Drug: Semuloparin sodium — 0.4 mL (0.2 mL if SRI) solution in ready-to-use 0.5 ml pre-filled syringe
  Subcutaneous injection once daily
  Other Names: AVE5026
  Arms: Semuloparin extension treatment

SUMMARY:
The primary objective is to evaluate the efficacy of once daily (QD) subcutaneous (SC) injections of Semuloparin sodium (AVE5026) versus placebo for 3 additional weeks following an initial 7 to 10-day venous thromboprophylaxis with open-label AVE5026 in patients having undergone hip fracture surgery.

The secondary objective is to evaluate the safety of extended AVE5026 administration.

DETAILED DESCRIPTION:
The total duration of observation per participant is 56-63 days from surgery broken down as follows:

* 7 to 10-day initial treatment period with open-label Semuloparin sodium;
* Randomization;
* 19 to 23-day double-blind treatment period with Semuloparin sodium or placebo;
* 30-day follow-up period.

Mandatory bilateral venography of the lower limbs is to be performed between 19 and 24 days after randomization.

ELIGIBILITY:
Inclusion Criteria:

* In the run-in phase:

  * Standard surgery for fracture of the upper third of the femur, including femoral head and neck
* In the double-blind phase following the run-in phase:

  * Completion of the run-in phase without permanent treatment discontinuation

Exclusion Criteria:

* Any major orthopedic surgery within 3 months prior to enrolment;
* Deep vein thrombosis or pulmonary embolism within the last 12 months, or known post-phlebitic syndrome;
* High risk of bleeding;
* Known hypersensitivity to heparins;
* Any contraindication to the performance of venography;
* End stage renal disease or patient on dialysis

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 469 (Actual)
Dates: Start 2008-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who Experience Venous Thromboembolism Events (VTE) or Death From Any Cause During the Extension Treatment Period | From randomization up to 24 days after randomization or the day of mandatory venography, whichever comes first
  VTE include any Deep Vein Thrombosis (DVT) (symptomatic or not) and non-fatal Pulmonary Embolism (PE) as confirmed by a Central Independent Adjudication Committee (CIAC) after review of mandatory bilateral venograms and diagnostic tests for suspected VTE. All-cause deaths include fatal PE and deaths for other reason than PE.

SECONDARY OUTCOMES:
Percentage of Participants Who Experience "Major" VTE or Death From Any Cause | From randomization up to 24 days after randomization or the day of mandatory venography, whichever comes first
  "Major" VTE include any proximal DVT, symptomatic distal DVT and non-fatal PE as confirmed by the CIAC.
Percentage of Participants Who Experience Clinically Relevant Bleedings During the Extension Treatment Period | From 1st study drug injection in the extension treatment period up to 3 days after last study drug injection
  Bleedings are centrally and blindly reviewed by the CIAC and classified as:
  "major" (fatal, in a critical area/organ, causing a post-operative drop in hemoglobin ≥2 g/dL or requiring post-operative transfusion ≥2 units of blood, leading to an invasive diagnostic or therapeutic intervention, or associated with circulatory decompensation);
  "clinically relevant non-major" (skin hematoma or epistaxis requiring surgical/medical intervention/treatment, macroscopic hematuria, or overt bleeding requiring specific attention by health care professional);
  "Non-clinically relevant bleeding".
Percentage of Participants Who Require the Initiation of Curative Anticoagulant or Thrombolytic Treatment After VTE Assessment During the Extension Treatment Period | From randomization up to 24 days after randomization or the day of mandatory venography, whichever comes first
  Initiation of curative anticoagulant or thrombolytic treatment after VTE assessment is defined from investigator's answer to the question "was the subject treated for VTE?" asked after the diagnostic tests for suspected VTE and after the mandatory venography.

OTHER OUTCOMES:
Overview of Reported Bleeding Adverse Event | From 1st study drug injection up to 3 days after last study drug injection
  Analysis periods are defined as follows:
  * Initial treatment: time from the first study drug injection up to the first injection in the extension period or up to 3 days after the last injection if no extension treatment;
  * Extension treatment: time from first injection in the extension period up to 3 days after the last injection.
Overview of Deaths | From 1st study drug injection up to 3 days after last study drug injection
  The same analysis periods as defined for the previous outcome measure are used. In addition deaths during the extension treatment period are centrally and blindly reviewed by the CIAC and classified as fatal PE, fatal bleeding, cardiovascular death or other based on relevant documentation (e.g. autopsy report).
Platelets Count: Percentage of Participants With Potentially Clinically Significant Abnormalities (PCSA) | From 1st study drug injection up to 3 days after last study drug injection
  PCSA are abnormal values considered medically important by the Sponsor according to pre-defined criteria based on literature review. Threshold for platelets count was defined as <100 Giga/L.
  The analysis periods as previously defined are used (see outcome measure 5).
Liver Function: Percentage of Participants With Potentially Clinically Significant Abnormalities (PCSA) | From 1st study drug injection up to 3 days after last study drug injection
  Thresholds are defined as follows:
  * Alanine Aminotransferase [ALT] >3 Upper Normal Limit [ULN];
  * Total Bilirubin [TB] >2 ULN;
  * ALT >3 ULN and TB >2 ULN;
  Cases with ALT >3 ULN and TB >2 ULN (not necessarily concomitant) are evaluated by a blinded independent adjudicator to determine if they met Hy's law criteria.
  The analysis periods as previously defined are used (see outcome measure 5).

CONTACTS AND LOCATIONS:
Overall Officials: William D. Fisher, MD, Principal Investigator — McGill University Health Centre, Montreal, Quebec, Canada; Alexander G. Turpie, MD, Study Chair — HHS-General Hospital, Hamilton, Ontario, Canada
Locations (16):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Minsk, Belarus
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Shangaï, China
- Sanofi-Aventis Administrative Office, Bogotá, Colombia
- Sanofi-Aventis Administrative Office, Cairo, Egypt
- Sanofi-Aventis Administrative Office, Mumbai, India
- Sanofi-Aventis Administrative Office, Vilnius, Lithuania
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Lima, Peru
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Midrand, South Africa
- Sanofi-Aventis Administrative Office, Seoul, South Korea
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)
- Sanofi-Aventis Administrative Office, Kiev, Ukraine

REFERENCES:
- [Result] Fisher WD, Agnelli G, George DJ, Kakkar AK, Lassen MR, Mismetti P, Mouret P, Turpie AG. Extended venous thromboembolism prophylaxis in patients undergoing hip fracture surgery - the SAVE-HIP3 study. Bone Joint J. 2013 Apr;95-B(4):459-66. doi: 10.1302/0301-620X.95B4.30730. PMID 23539696